CLINICAL TRIAL: NCT05181293
Title: Impact of a Mobile Gaming App on Infant and Young Child Feeding Practices of Teenage Mothers, and Nutritional Status of Children (0 - 24 Months) in Nigeria
Brief Title: Mobile Gaming App to Improve Child Nutrition in Nigeria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Jeanne Freeland-Graves, The Bess Heflin Centennial Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00001047
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Child Malnutrition; Behavior, Maternal
MeSH Terms: conditions — Child Nutrition Disorders; Behavior | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): A mobile gaming app (BabyThrive) will be disseminated to teenage mothers to help them learn about exclusive breastfeeding, introduction to solid/semi-solid foods, meal frequency and dietary diversity. BabyThrive will also demonstrate how to prepare 30 nutritious recipes for complementary feeding; create a calendar and set reminders to prompt mothers to access child health services; and plot growth patterns of the baby to facilitate growth monitoring.
  Interventions: Behavioral: Mobile Gaming App for Nutrition Intervention
- No Intervention (No Intervention): In addition to routine health services, teenage mothers will receive the BabyThrive app after the intervention is completed. Participants will learn about exclusive breastfeeding, introduction to solid/semi-solid foods, meal frequency and dietary diversity. BabyThrive also will demonstrate how to prepare 30 nutritious recipes for complementary feeding; create a calendar and set reminders to prompt mothers to access child health services; and plot growth patterns of baby to facilitate growth monitoring.

INTERVENTIONS:
Behavioral: Mobile Gaming App for Nutrition Intervention — A mobile gaming app (BabyThrive) will be disseminated to teenage mothers to help them learn about exclusive breastfeeding, introduction to solid/semi-solid foods, meal frequency and dietary diversity. BabyThrive will also demonstrate how to prepare 30 nutritious recipes for complementary feeding; create a calendar and set reminders to prompt mothers to access child health services; and plot growth patterns of the baby to facilitate growth monitoring.
  Arms: Experimental

SUMMARY:
Undernutrition among children born to teenage mothers deserves urgent attention in Nigeria, where 27.2% of girls (15-19 years) living in rural areas have begun childbearing. The overall goal of this study is to develop, validate and evaluate the effects of a mobile gaming app on the infant and young child feeding practices of teenage mothers, and the nutritional status of children (0 - 2 years).

DETAILED DESCRIPTION:
Undernutrition among children born to teenage mothers deserves urgent attention in Nigeria, where 27.2% of girls (15-19 years) living in rural areas have begun childbearing. Pregnancy elevates the nutrient needs of teenage girls due to competing requirements for fetal development, and growth and maturity in the adolescent mother. The resultant children have a higher likelihood of underweight (13-fold), stunting (8-fold) and wasting (3-fold), and are over 50% more likely to die within the first month of birth, as compared to children of older mothers. Previous studies have found positive associations between maternal education/knowledge and optimum infant and young child feeding (IYCF) practices. Childbirth results in a sharp increase in the responsibilities and work burden of teenage mothers, negatively impacting capacity and self-efficacy for adequate child feeding. Furthermore, attempts to improve IYCF practices often target older women. The overall goal of this study is to develop, validate and evaluate the effects of a mobile gaming app on the infant and young child feeding practices of teenage mothers. A secondary goal is to evaluate the anthropometric and dietary and plasma levels of microminerals of children, 0 - 24 months of age. A mobile app will be developed and validated. It will feature an interactive role-play game on recommended IYCF practices that will help educate teenage mothers about feeding young children. A 6-month randomized controlled trial (RCT) will be conducted in 266 predominantly low-income mother-child dyads (0 - 24 months) from Nigeria. This RCT will compare the influence of the BabyThrive app vs controls who receive a delayed intervention. It will include knowledge and practices regarding exclusive breastfeeding, introduction to solid/semi-solid foods, meal frequency, dietary diversity and amount of food consumed of teenage mothers. Anthropometric measurements and plasma ferritin and zinc of children also will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Teenage mothers with children aged 0 - 24 months

Exclusion Criteria:

* Children with acute infections, metabolic or feeding issues
* Mothers younger than 14 years of age
* HIV-positive mothers

Ages: 0 Months to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 216 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Infant and Young Child Feeding (IYCF) knowledge and practice scores of teenage mothers | Baseline, Month 6 of intervention
  Mean change in scores from baseline, after 6 months of intervention. Measured at baseline and at 6 months after the intervention, using the Teen Moms IYCF Questionnaire (to be validated at the beginning of this study)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne H Freeland-Graves, PhD, RD, Principal Investigator — University of Texas at Austin
Locations (1):
- Center for Family Health Initiative, Abuja, Federal Capital Territory, Nigeria

IPD SHARING:
Plan to Share IPD: No